CLINICAL TRIAL: NCT01253707
Title: A Phase 1, First-In-Human Study Evaluating the Safety, Tolerability, and Pharmacokinetics of AMG 337 in Adult Subjects With Advanced Solid Tumors
Brief Title: A Study of AMG 337 in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20101132
Record Dates: First submitted 2010-11-24; First posted 2010-12-03 (Estimated); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Advanced Malignancy; Advanced Solid Tumors; Cancer; Oncology; Oncology Patients; Tumors
Keywords: Solid Tumors; C-met inhibitor
MeSH Terms: conditions — Neoplasms | interventions — AMG 337

ARMS (1):
- Dose Escalation (Experimental)
  Interventions: Drug: AMG 337

INTERVENTIONS:
Drug: AMG 337 — AMG 337 is a small molecule inhibitor of c-Met which is a receptor tyrosine kinase expressed on the surface of epithelial cells.

SUMMARY:
First in human, open-label, sequential dose escalation and expansion study of AMG 337 in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 18 years old
* Subjects must have a pathologically documented, definitively diagnosed, advanced solid tumor
* Subjects with primary central nervous system (CNS) tumors or metastases resected or have received radiation therapy ending at least 4 weeks prior to study day 1 are eligible providing they meet all of the following criteria: a) residual neurological symptoms grade ≤ 1; 2) no dexamethasone treatment; and c) follow-up MRI shows no new lesions appearing
* Measurable disease per RECIST guidelines (subjects with non-measurable, but evaluable disease are also eligible for the dose escalation portion of the study)
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2
* Competent to sign and date an Institutional Review Board approved informed consent form
* Adequate hematologic and renal function as determined by laboratory blood and urine tests

Exclusion Criteria:

* Men and woman of reproductive potential, unwilling to practice a highly effective method of birth control for the duration of the study and continuing for 2 weeks (for women) and 12 weeks (for men) after receiving the last dose of study drug.
* Women who are lactating/breastfeeding or planning to become pregnant during the duration of the study
* History of bleeding diathesis
* Myocardial infarction within 6 months of study day 1, symptomatic congestive heart failure (New York Heart Association > class II), unstable angina, or unstable cardiac arrhythmia requiring medication, or uncontrolled hypertension
* A baseline ECG QTc > 470 ms
* Active infection requiring (IV) antibiotics within 2 weeks of study enrollment
* Significant gastrointestinal disorder(s), in the opinion of the investigator, that may influence drug absorption
* Known positive test for HIV
* Known acute or chronic hepatitis B or hepatitis C infection as determined by serologic tests
* Anti-tumor therapy within 28 days of study day 1 including chemotherapy, antibody therapy, retinoid therapy, or other investigational agent
* Major surgery within 30 days of study day 1
* Any co-morbid medical disorder that may increase the risk of toxicity, in the opinion of the investigator or sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2010-12-08 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2016-12-13 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of AMG 337 by reviewing clinically significant or ≥ Grade 3 changes in safety laboratory tests, physical examinations, ECGs, or vitals signs in all subjects enrolled. | 4 years
Characterize the pharmacokinetics of AMG 337 when administered orally. PK parameters will include, but are not limited to, area under the plasma concentration versus time curve (AUC) and Peak Plasma Concentration (Cmax). | 4 years
Determine the maximum tolerated dose of AMG 337, if possible. The MTD is defined at the highest dose level with an observed incidence of dose limiting toxicity in < 33% of subjects enrolled in a cohort. | 4 years

SECONDARY OUTCOMES:
Evaluate for clinical responses associated with AMG 337 treatment according to Response Evaluation Criteria In Solid Tumors 1.1 criteria | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (8):
- United States (8):
  - Research Site, Los Angeles, California
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Columbus, Ohio
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas

REFERENCES:
- [Background] Amouzadeh HR, Dimery I, Werner J, Ngarmchamnanrith G, Engwall MJ, Vargas HM, Arrindell D. Clinical Implications and Translation of an Off-Target Pharmacology Profiling Hit: Adenosine Uptake Inhibition In Vitro. Transl Oncol. 2019 Oct;12(10):1296-1304. doi: 10.1016/j.tranon.2019.05.018. Epub 2019 Jul 19. PMID 31330495
- [Background] Hong DS, LoRusso P, Hamid O, Janku F, Kittaneh M, Catenacci DVT, Chan E, Bekaii-Saab T, Gadgeel SM, Loberg RD, Amore BM, Hwang YC, Tang R, Ngarmchamnanrith G, Kwak EL. Phase I Study of AMG 337, a Highly Selective Small-molecule MET Inhibitor, in Patients with Advanced Solid Tumors. Clin Cancer Res. 2019 Apr 15;25(8):2403-2413. doi: 10.1158/1078-0432.CCR-18-1341. Epub 2018 Nov 13. PMID 30425090
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com